CLINICAL TRIAL: NCT00489463
Title: The Effect of the Levonorgestrel-Releasing Intrauterine System and the Copper-Intrauterine Device (TCu 380A) on Subendometrial Microvascularization and Uterine Artery Blood Flow.
Brief Title: IUD Uterine Vascularization and Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IUD vascularization
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2006-01

CONDITIONS: Healthy
Keywords: LNG-IUS; TCu 380A; Ultrasonography; Doppler color; power Doppler; female; Volunteers
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: intra-uterine device (TCu 380A)

SUMMARY:
The aim of this study was to evaluate the effect of the LNG-IUS and TCU 380A users on the sub-endometrial vascularization and the uterine artery blood flow using power Doppler analysis and ultrasonography pulsed color Doppler during the precise mid-luteal phase.

DETAILED DESCRIPTION:
Design We will perform a prospective (quasi-experimental) clinical trial. Patients/Methodology We prospectively will enrolled consecutive patients who wants to use IUD (LNG-IUS or TCU 380A). We will evaluate the sub-endometrial blood flow using power Doppler analysis, uterine artery blood flow using pulsatility and resistance index and endometrial thickness before IUD insertion and three months later.

The inclusion criteria are: 1. regularly menstruating women (menstrual cycle varying between 24-35 days); 2. Normal serum TSH, FSH and prolactin levels (as measured on day-3) and with less than 40 years. Contraceptive pills or any kind of hormonal medication had not been taken for (at least) 3 months prior to the study and any intrauterine device had necessarily been removed at least 3 months earlier. Patients will be allowed to not use non-steroidal anti-inflammatory drugs (NSAID) within 24 h prior to any examination.

The exclusion criteria are pregnancy, acute or chronic pelvic inflammatory disease, menorrhagia for unknown reason, copper allergy, cervicitis, dysplasia in the cervix or genital tumor. All patients underwent a gynecological examination and had a Papanicolaou smear taken during the previous 12 months.

All patients will be daily examined with US after the eighth day of the cycle, and follicular development will be observed to confirm ovulation; they are then examined in the mid-luteal phase, 6-9 days after ovulation, to obtain the power Doppler energy (PDE) measurement, pulsatility index (PI), resistance index (RI) and endometrial thickness (ET) by ultrasound (US) scans. The study was approved by the Ethical Committee of Hospital de Clinicas de Porto Alegre, IRB equivalent (# 02-127) and informed consent was obtained from all patients.

Patients will be allocated into 2 groups according to the IUD: LNG-IUS (group A) or TCu 380A (group B).

Three months after the LNG-IUS (group A) or TCu 380A (group B) insertion, also in the mid-luteal phase (6-9 days after ovulation, confirmed by US), all subjects repeated the same study protocol.

The sonographic equipment that will be used consisted of a SONOACE 9900 (Medison SA - Korea). The PDE, PI and RI will be performed on a transvaginal route. The settings for Power Doppler sonography are standardized for the highest sensitivity in the absence of apparent noise using a high pass filter at 50 Hz, pulsed repetition frequency at 750 Hz, and moderate long persistence. The lowest possible measurable velocity was below 5 cm/s. The same investigator, using the same equipment and parameters will performe the sonography assessments so as to eliminate any interobserver variation. All exams were carried out between 08:00 and 10:00 a.m. in order to avoid interference of the circadian rhythm (10).

Power Doppler energy is classified into 5 categories according to the sub-endometrial signal area percentage: I (<10%), II (10-25%), III (25-50%), IV (50-75%) and V (>75%).

Statistics Student t test is used for comparing age and body mass index (BMI). The Wilcoxon-Mann-Whitney (WMW) test is used to compare skewed data (PI, RI and ET), whereas the Chi-Square test and Fisher's exact test are used for categorical data (PDE).

We will use multiple logistic regression model to examine the association of the outcome (PI variability, before and after IUD insertion), categorized in percentile 50 and IUD (LNG-IUS or TCu 380A), age (years), and parity (0,1 or >1) the independent variables. P-value < 0.05 was considered statistically significant. The power calculation before this study protocol required the inclusion of 19 patients for a Pß=80%.

ELIGIBILITY:
Inclusion Criteria:

* Regularly menstruating women (menstrual cycle varying between 24-35 days);
* Normal serum TSH, FSH and prolactin levels (as measured on day-3) and with less than 40 years. Contraceptive pills or any kind of hormonal medication had not been taken for (at least) 3 months prior to the study and any intrauterine device had necessarily been removed at least 3 months earlier. Patients were allowed to not use non-steroidal anti-inflammatory drugs (NSAID) within 24 h prior to any examination.

Exclusion Criteria:

* Pregnancy, acute or chronic pelvic inflammatory disease, menorrhagia for unknown reason, copper allergy, cervicitis, dysplasia in the cervix or genital tumor. All patients underwent a gynecological examination and had a Papanicolaou smear taken during the previous 12 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2004-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Ultra-sound doppler, IP and IR indexes | 3 mo

SECONDARY OUTCOMES:
pelvic pain, uterine bleediing | 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: Joao Cunha-Filho, PhD, Principal Investigator — Professor UFRGS
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, RGS, Brazil